CLINICAL TRIAL: NCT01174628
Title: The ELOPE Study: Prospective Evaluation of Long-term Outcomes After Pulmonary Embolism
Brief Title: Prospective Evaluation of Long-term Outcomes After Pulmonary Embolism
Acronym: ELOPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Susan Kahn, M.D., M.Sc., Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: MOP-93627
Record Dates: First submitted 2010-07-28; First posted 2010-08-03 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Pulmonary Embolism
Keywords: Exercise Tolerance; Venous Thrombosis; Pulmonary Embolism; Quality of Life (QOL)
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — platelet-poor plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the long-term impact of Pulmonary Embolism (PE) on heart and lung function, quality of life, ability to work, symptoms of breathlessness and functional status of patients one year after their initial diagnosis and treatment for PE

ELIGIBILITY:
Inclusion Criteria:

1. First episode of acute symptomatic PE that was objectively diagnosed* within last 10 days
2. Treated with anticoagulants
3. ≥ 18 years old

   * PE will be diagnosed if there is a high probability V/Q scan (as per PIOPED Study criteria 66), an intraluminal filling defect in segmental or larger vessels on CTPA or a constant intraluminal filling defect or abrupt cut-off of vessels greater than 2.5 mm diameter on pulmonary angiography 8,10. Patients with non-definitive test results (e.g. low or intermediate probability V/Q scan, subsegmental PE on CTPA (~5% of PE patients 12) will not be included in order to have a strictly defined population of patients with definite PE.

Exclusion Criteria:

1. Contraindication or unable to perform CPET or 6MWT (amputated or paralyzed limb(s), severe lower extremity arthritis, preexisting cardiopulmonary condition precluding exercise including unstable angina or myocardial infarction in last 6 weeks, uncontrolled hypertension, serious cardiac dysrhythmia on resting EKG [severe bradycardia or tachycardia, sick sinus syndrome or multifocal premature ventricular contractions] and syncope)
2. Contraindication to CTPA (allergy to iodinated contrast, CrCl or eGFR < 30 ml/min)
3. Severe comorbidity (congestive heart failure [LVEF < 35%], severe COPD or restrictive lung disease [FEV1<50%, chronic need for oxygen therapy])
4. Previous DVT (as ~40% of patients with proximal DVT have asymptomatic PE on lung imaging 67)
5. Life expectancy < 1 year (e.g. active or terminal cancer, end-stage cardiac or respiratory disease).
6. Pregnancy or lactation
7. Unable to read questionnaire in English or French
8. Unable to return to study centre for required follow-up visits
9. Unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the Emergency Department, in-patient wards, out-patient clinics or anticoagulation clinics.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Exercise Limitation | 1 month
  Exercise limitation will be assessed by VO2 max (% predicted) on cardiopulmonary exercise testing (CPET)
Exercise Limitation | 12 months
  Exercise limitation will be assessed by VO2 max (% predicted) on cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Quality of Life | Baseline
  Quality of Life will be assessed using the SF-36v2 questionnaire.
Quality of Life | 1 month
  Quality of Life will be assessed using the SF-36v2 questionnaire.
Quality of Life | 3 months
  Quality of Life will be assessed using the SF-36v2 questionnaire.
Quality of Life | 6 months
  Quality of Life will be assessed using the SF-36v2 questionnaire.
Quality of Life | 12 months
  Quality of Life will be assessed using the SF-36v2 questionnaire.
Respiratory Disease-Specific Measures | Baseline
  Respiratory Disease-Specific measures will be assessed using the Pulmonary Embolism Quality of Life Questionnaire (PEmb-QOL) and the San Diego Shortness of Breath Questionnaire (SOBQ).
Respiratory Disease-Specific Measures | 1 month
  Respiratory Disease-Specific measures will be assessed using the Pulmonary Embolism Quality of Life Questionnaire (PEmb-QOL) and the San Diego Shortness of Breath Questionnaire (SOBQ).
Respiratory Disease-Specific Measures | 3 months
  Respiratory Disease-Specific measures will be assessed using the Pulmonary Embolism Quality of Life Questionnaire (PEmb-QOL) and the San Diego Shortness of Breath Questionnaire (SOBQ).
Respiratory Disease-Specific Measures | 6 months
  Respiratory Disease-Specific measures will be assessed using the Pulmonary Embolism Quality of Life Questionnaire (PEmb-QOL) and the San Diego Shortness of Breath Questionnaire (SOBQ).
Respiratory Disease-Specific Measures | 12 months
  Respiratory Disease-Specific measures will be assessed using the Pulmonary Embolism Quality of Life Questionnaire (PEmb-QOL) and the San Diego Shortness of Breath Questionnaire (SOBQ).

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Kahn, M.D., M.Sc., Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital; Andrew Hirsch, M.D., Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital; John Granton, M.D., Principal Investigator — University of Toronto
Locations (5):
- Canada (5):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec

REFERENCES:
- [Derived] Kahn SR, Hirsch AM, Akaberi A, Hernandez P, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Geerts WH, Aaron SD, Granton JT. Functional and Exercise Limitations After a First Episode of Pulmonary Embolism: Results of the ELOPE Prospective Cohort Study. Chest. 2017 May;151(5):1058-1068. doi: 10.1016/j.chest.2016.11.030. Epub 2016 Dec 6. PMID 27932051
- [Derived] Kahn SR, Houweling AH, Granton J, Rudski L, Dennie C, Hirsch A. Long-term outcomes after pulmonary embolism: current knowledge and future research. Blood Coagul Fibrinolysis. 2014 Jul;25(5):407-15. doi: 10.1097/MBC.0000000000000070. PMID 24469387